CLINICAL TRIAL: NCT05627401
Title: Customized Modified Multiple Orbital Wall Decompression With Fat Removal for Sight-threatening Graves's Ophthalmopathy : a Retrospective Cohort Study
Brief Title: Customized Multiple Orbital Wall Decompression for Sight-threatening Graves's Ophthalmopathy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Other Study IDs: SYSKY-2022-349-01
Record Dates: First submitted 2022-11-17; First posted 2022-11-25 (Actual); Last update posted 2022-11-25 (Actual); Status verified 2022-11

CONDITIONS: Thyroid Eye Disease
Keywords: Orbital decompression; Graves' orbitopathy; Dysthyroid optic neuropathy
MeSH Terms: conditions — Graves Ophthalmopathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Single Group Assignment: patients with sight-threatening Graves orbitopathy (GO) who underwent customized/individual multiple orbital wall decompression plus fat removal
  Interventions: Procedure: Modified multiple orbital wall decompression

INTERVENTIONS:
Procedure: Modified multiple orbital wall decompression — Thyroid dysfunction of all patients is stabilized by ATDs until treatment of TAO is completed. All patients with sight-threatening GO were admitted for emergency steroid pulse therapy. And additional drugs for protecting gastrointestinal mucous membrane, potassium and calcium supplements, and sedatives were used. All emergency cases, whose signs of visual impairment clinically attributable to GO existed despite first-line steroid treatment, were referred and discussed at the surgical board of our interdisciplinary center for prompt surgical orbital decompression. Urgent orbital decompression was performed when response is absent or poor within 1-2 weeks.

SUMMARY:
Graves' orbitopathy (GO) is an disfiguring and disabling autoimmune condition. Sight-threatening GO is an most severe form and occurs in about 5% of patients with Graves' disease. It can cause blurred vision, color vision and vision function damage, and affects the quality of life. The goal of this retrospective cohort study is to propose a customized orbital decompression algorithm for patients with sight-threatening Graves'ophthalmopathy and to explore the therapeutic effect of customized orbital decompression in sight-threatening patients.

ELIGIBILITY:
Inclusion Criteria:

* Sight-threatening patients undergoing interdisciplinary discussion and orbital decompression operation.
* The sight-threatening GO refer to those with DON, exposure keratitis or corneal breakdown.
* DON was diagnosed according to the following clinical findings including optic nerve head edema, visual field defect, impaired color vision, afferent pupil defect, retinal folds, radiologic evidence of apical optic nerve compression or globe subluxation.
* Diagnosis of exposure keratitis or corneal breakdown was made based on physical exam signs, e.g. microepithelial defects, abrasion or ulcer. A minimum follow-up of 12 months was required for inclusion.

Exclusion Criteria:

* Patients were excluded if exophthalmos, rather than acute visual loss, was the indication for surgery.
* Cases with a history of previous ocular surgery, glaucoma, and visual defects from other ocular conditions were excluded from the study.

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: This was a retrospective cohort study of patients with sight-threatening Graves orbitopathy (GO) who underwent customized/individual multiple orbital wall decompression plus fat removal at Sun Yat-Sen Memorial Hospital from Jan. 2017 to Dec. 2021.
Sampling Method: Probability Sample
Enrollment: 78 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
BCVA | 12 months
  best corrected visual acuity in logMAR
CAS | 12 months
  clinical activity score
proptosis | 12 months
  proptosis in mm
EVP | 12 months
  Visual Evoked Potential

SECONDARY OUTCOMES:
GO-QOL | 12 months
  Graves' Ophthalmopathy Quality of Life

CONTACTS AND LOCATIONS:
Overall Officials: Peng Tian, PhD., M.D., Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen Memorial Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No
Medical records or outpatient examination records cannot be shared by hospitals across the country.

REFERENCES:
- [Derived] Tian P, Zeng P, Zhang H, Liang J, Li E, Ma Y, Zou H, Wang M, Xiang L. Balanced medial-lateral wall vs selective 3-wall orbital decompression for sight-threatening Graves's orbitopathy: a clinical retrospective cohort study from 2016 to 2022. Eur Arch Otorhinolaryngol. 2024 Sep;281(9):4807-4815. doi: 10.1007/s00405-024-08589-x. Epub 2024 Apr 13. PMID 38613579